CLINICAL TRIAL: NCT06439420
Title: Cognitive Behavioral Therapy for Insomnia in Brain Tumor Patients: Phase IIc Randomized Feasibility Pilot Trial
Brief Title: CBT-I in Primary Brain Tumor Patients: Phase IIc Randomized Feasibility Pilot Trial
Acronym: CBT-I in PBT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-23-20323; HM20028336 (Other: Virginia Commonwealth University)
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Primary Brain Tumor; Glioblastoma; Astrocytoma; Oligodendroglioma; Meningioma; Primary Central Nervous System (CNS) Lymphoma
Keywords: Brain Tumor; Insomnia; Glioma; Sleep
MeSH Terms: conditions — Brain Neoplasms; Glioblastoma; Astrocytoma; Oligodendroglioma; Meningioma; Lymphoma; Sleep Initiation and Maintenance Disorders; Glioma | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth Cognitive Behavioral Therapy for Insomnia (Experimental)
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia
- Enhanced Treatment as Usual (No Intervention)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia — CBT-I is a non-pharmacological approach to treating sleep disturbance consisting of educational, behavioral, and cognitive intervention components with evidence-based strategies including sleep efficiency, stimulus control, and sleep hygiene modification. CBT-I includes at least 6 group sessions, each approximately 90 minutes in length, delivered over 6 weeks via telehealth.
  Arms: Telehealth Cognitive Behavioral Therapy for Insomnia

SUMMARY:
This study seeks to investigate an evidence-based, manualized, behavioral health intervention, Cognitive Behavioral Therapy for Insomnia (CBT-I), in individuals with primary brain tumors (PBT) and insomnia. Our project will assess the feasibility and acceptability of recruitment, enrollment, data collection procedures, and retention of individuals with PBT and insomnia in the behavioral health intervention, CBT-I, and investigate the potential benefits of CBT-I within this at-risk and understudied population. In the long term, the goals are to expand treatment options for neuro-oncology patients and improve their mission readiness and overall wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* Primary brain tumor diagnosis (grade I-IV)
* >/=2weeks post-cranial resection (if applicable)
* >/=1 month post-radiation therapy (if applicable)
* Able to understand, speak, and read English
* Absence of major cognitive concerns
* Meet Diagnostic and statistical manual of mental disorders version 5 (DSM-V) diagnostic criteria for insomnia
* Reliable internet connection

Exclusion Criteria:

* Major communication difficulties that would prohibit effective intervention
* Inability to attend weekly virtual group meetings
* Inability to understand and provide informed consent
* Currently a prisoner or residing in a correctional facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-07-08 (Actual); Primary Completion 2025-09-25 (Actual); Study Completion 2025-09-25 (Actual)

PRIMARY OUTCOMES:
Rate of consent to screening procedures | Baseline (Day 1)
  Number of participants that consent to screening procedures
Rate of those eligible enrolling | Baseline (Day 1)
  Number of participants that are eligible to enroll to the protocol
Rate of baseline assessment completion | Week 1
  Number of participants that complete the baseline assessment
Rate of post-intervention assessment completion | Week 6
  The number of participants that complete the post-intervention assessment
Rate of follow-up assessment completion | Week 18
  The number of participants that complete the follow-up assessment
Rate of intervention attrition | Week 6
  The number of participants that do not complete the CBT-I intervention
Acceptability of quantity of assessments | Week 18
  Satisfaction rating of quantity of assessments on a scale of 1-5 with 5 being the best
Acceptability of timing of assessments | Week 18
  Satisfaction ratings of timing of assessments on a scale of 1-5 with 5 being the best
Acceptability of duration of assessments | Week 18
  Satisfaction ratings of duration of assessments on a scale of 1-5 with 5 being the best

CONTACTS AND LOCATIONS:
Overall Officials: Ashlee Loughan, Ph.D, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data.